CLINICAL TRIAL: NCT05462041
Title: Evaluating the Safety of Utilizing Donor Hearts From Donation After Circulatory Death (DCD) Donors Compared to Donor Hearts From Donation After Brain Death (DBD) Donors: A Single Center Pilot Study
Brief Title: DCD IIT: Evaluating the Safety of Utilizing Donor Hearts From Donation After Circulatory Death (DCD) Donors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Fardad Esmailian, Surgical Director, Heart Transplantation and Mechanical Circulatory Support, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00002090
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Organ Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- DBD Donor Heart Transplantation (Other): If the heart offer is from a DBD donor, the heart will be retrieved per standard of care.
  Interventions: Other: DBD Donor Heart Transplantation
- DCD Donor Heart Transplantation (Other): If the heart offer is from a DCD donor, the heart will be retrieved using one of two strategies: Normothermic Regional Perfusion (NRP) or Direct Procurement and Perfusion (DPP). NRP procedures will be used to procure all DCD hearts unless contraindicated or prohibited by the donor hospital. In the event the donor hospital does not allow NRP for cardiac organ procurement, or the target number of eight DCD transplants with NRP has been achieved, DPP with the Organ Care System (OCS) should be utilized.
  Interventions: Device: DCD Donor Heart Transplantation

INTERVENTIONS:
Other: DBD Donor Heart Transplantation — A technique of donor heart procurement.
  Arms: DBD Donor Heart Transplantation
Device: DCD Donor Heart Transplantation — A technique of donor heart procurement. The TransMedics' OCS Heart technology is the only portable system available for ex-vivo maintenance of the donor heart in a metabolically active and beating state. It is currently FDA approved for procurement and transport.
  Arms: DCD Donor Heart Transplantation

SUMMARY:
The purpose the research is to evaluate whether patients who receive a Donation after Circulatory Death (DCD) heart for cardiac transplantation using either normothermic regional perfusion (NRP) or direct procurement and perfusion (DPP) have similar outcomes as patients who receive Donation after Brain Death (DBD) heart using standard cold storage. The study will also evaluate whether DCD procured hearts have a meaningful impact on hearts available for transplantation at our center.

DETAILED DESCRIPTION:
In the U.S., heart donation occurs after a person has been declared brain dead and is called a donor after brain death (DBD). In these patients, the heart continues to beat and pump blood throughout the body. After life support is withdrawn, organs are retrieved immediately for transplantation. This study will use hearts from donors after circulatory death (DCD) donors. DCD donors are those whose hearts have stopped beating and no longer pump blood. DCD hearts are not used as often for transplantation today in the U.S. because they may be further injured during traditional cold storage. In the US, donor hearts are currently mostly obtained from donors after brain death (DBD), although DCD donors are used for other donated organs, such as: lungs, kidneys, and livers.

This study will evaluate whether patients who receive a DCD heart transplant using either NRP or DPP have similar outcomes as patients who receive DBD hearts using standard cold storage. The study will also evaluate whether DCD procured hearts have a meaningful impact on hearts available for transplantation at our center. Ten (10) DCD donor heart recipients will be enrolled into the study intervention group, and approximately 30 DBD donor heart recipients will be enrolled into the control group.

ELIGIBILITY:
Recipient Inclusion Criteria:

1. Subjects must be willing and be capable of understanding the purpose and risks of the study and must sign a statement of informed consent OR consent of a legally authorized representative of a cognitively impaired individual will be obtained before the cognitively impaired individual may be included in research.
2. Signed: 1) written informed consent document and 2) authorization to use and disclose protected health information
3. Male or female, aged 18 years of age or older listed for primary heart transplant

Recipient Exclusion Criteria:

1. Prior history of cardiac transplantation
2. Multi-organ transplant
3. Current or planned participation in another interventional trial
4. Recipient has any condition that, in the opinion of the Investigator, would make study participation unsafe or would interfere with the objectives of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of utilizing DCD donor hearts as compared to DBD donor hearts for transplantation. | 30 days post-heart transplant
  Percentage of subjects with incidence of heart graft-related Serious Adverse Events (HGRSAEs) in the DCD Heart Transplanted Recipient Population

SECONDARY OUTCOMES:
Assess the practical, financial and logistical viability of using NRP vs. DPP for the procurement of DCD donor hearts. | 1 year
  Length of time on waiting list for DCD hearts (compared to time on waiting list for DBD heart for that patient, and compared to the median time for a patient matched for height and ABO group)

CONTACTS AND LOCATIONS:
Overall Officials: Fardad Esmailian, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

DOCUMENTS (1):
  • Study Protocol (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT05462041/Prot_001.pdf